CLINICAL TRIAL: NCT04594720
Title: Using Circulating Biomarkers to Identify Thyroid Cancer From the Patients With Thyroid Nodules
Brief Title: Circulating Biomarkers to Identify Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801437B0
Record Dates: First submitted 2020-10-16; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Thyroid Cancer; Thyroid Cancer, Papillary; Benign Thyroid Tumor
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid cancers: Enrolled study population have papillary thyroid cancers and benign thyroid tumors
  Interventions: Other: Identification group; Other: Validation group

INTERVENTIONS:
Other: Identification group — papillary thyroid cancers (n=10) and benign thyroid tumors (n=10)
Other: Validation group — papillary thyroid cancers (n=45) and benign thyroid tumors (n=35)

SUMMARY:
This study aimed to identify the potential circulating biomarkers of protein, mRNAs, and long non-coding RNAs (lncRNAs) to diﬀerentiate the papillary thyroid cancers from benign thyroid tumors. Methods: The study population of 100 patients was classified into identification (10 patients with papillary thyroid cancers and 10 patients with benign thyroid tumors) and validation groups (45 patients with papillary thyroid cancers and 35 patients with benign thyroid tumors). The Sengenics Immunome Protein Array combined data mining approach using the Open Targets Platform was used to identify the putative protein biomarkers, and their expression validated using the enzyme-linked immunosorbent assay. Next-generation sequencing by Illumina HiSeq was used for the detection of dysregulated mRNAs and lncRNAs. The website Timer v2.0 helped identify the putative mRNA biomarkers, which were significantly over-expressed in papillary thyroid cancers than in adjacent normal thyroid tissue. The mRNA and lncRNAs biomarker expression was validated by a real-time polymerase chain reaction.

DETAILED DESCRIPTION:
Novel biomarkers identification from liquid biopsy samples is in great demand for the diagnosis for malignant diseases. Generally, blood sampling is less invasive and could be carried out repeatedly. In addition to protein markers, circulating nucleic acids are promising sources of cancer biomarkers , since circulating nucleic acids provide information on the genome or gene expression , and harbor wealth of health and disease status information. The long non-coding RNAs (lncRNAs) are the transcripts longer than 200 nucleotides in length and act as prominent regulators of gene expression. Accumulating evidence demonstrated the involvement of lncRNA dysregulation in a variety of cancers, and their expression is associated with cancer development and metastasis. This study was designed to identify the potential protein and RNA biomarkers in the blood for diﬀerentiating a malignant thyroid tumor from a benign thyroid nodule. In this study, only patients with papillary thyroid carcinoma, the most common type of thyroid cancer, were chosen for comparison with those with benign thyroid tumors to simplify the comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid nodules who received total or subtotal thyroidectomy
* Patients aged 20 years and above

Exclusion Criteria:

* Patients with any other type of cancer, immunocompromised disease, or autoimmune disease.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was assigned to identification (10 patients with papillary thyroid cancers and 10 patients with benign thyroid tumors) and validation groups (45 patients with papillary thyroid cancers and 35 patients with benign thyroid tumors). Before surgery, 2 mL blood samples were drawn from an elbow vein of patients into EDTA tubes (BD Vacutainer) for RNA analysis, and 8 mL into SST™II advance tubes (BD Vacutainer) for protein analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Stage of thyroid cancers | 1 months after surgery
  The final diagnosis of malignant or benign lesions was based on the pathological reports.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan